CLINICAL TRIAL: NCT03533738
Title: Effects of Food Sequence on the Glycaemic and Insulinaemic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/00742
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Food selection 1 (Experimental): To consume vegetables followed by meat & rice together
  Interventions: Other: Food sequence 1
- Food selection 2 (Experimental): To consume meat followed by vegetables & rice together
  Interventions: Other: Food sequence 2
- Food selection 3 (Experimental): To consume as follows: vegetables, meat, rice
  Interventions: Other: Food sequence 3
- Food selection 4 (Experimental): To consume vegetables followed by meat and rice together
  Interventions: Other: Food sequence 4
- Food selection 5 (Experimental): To consume rice followed by vegetables & meat together
  Interventions: Other: Food sequence 5

INTERVENTIONS:
Other: Food sequence 1 — Vegetables first then meat & rice together
  Arms: Food selection 1
Other: Food sequence 2 — Meat first then vegetables & rice together
  Arms: Food selection 2
Other: Food sequence 3 — Vegetables first then meat followed by rice
  Arms: Food selection 3
Other: Food sequence 4 — Vegetables first followed by meat and rice together
  Arms: Food selection 4
Other: Food sequence 5 — Rice first followed by vegetables & meat together
  Arms: Food selection 5

SUMMARY:
The study hypothesizes that vegetable and protein consumed before a carbohydrate will reduce the glucose response. The vegetables and protein consumed before carbohydrate have different effects on insulin and satiety responses.

DETAILED DESCRIPTION:
Up to 20 healthy subjects will be recruited for the study and before inclusion in the study, potential participants will be given the opportunity to ask questions. Subjects who will fulfill all the acceptable criteria(Chinese ethnicity, body mass index between 18-25 kg/m2, weight of at least 45kg, normal blood pressure,less than or equal 140 and 90 mmHg; age between 21-40 years, fasting blood glucose less than 6 mmol/L) may be included in the study.Each subject will be asked to complete a screening session(lasting approximately1 hour) in a fasted state where baseline measurements including anthropometric measurements, fasting blood glucose and blood pressure will be collected from each participant to assess their eligibility.On the day before each test, enrolled subjects will be asked to restrict their intake of alcohol and caffeine-containing drinks and to restrict their participation in intense physical activity (eg, long periods at the gym, intensive swimming, running, aerobics etc). There is a total of five test sessions. Test sessions will be interspaced by a minimum of 1 week. For each session, subjects are required to come between 8:00-9:00am, with each session lasting approximately 4 hours. Subjects would have to come following a 10-12 hour overnight fast. An indwelling catheter will be inserted into a vein in your forearm and will be kept patent (free of clots) for the remainder of the test session. The investigators will then take a blood sample from the cannula to measure baseline values. The investigators will also take a finger prick blood sample to measure blood glucose concentration. After obtaining the baseline blood samples the investigators will give subjects the test meal in different sequence consume in 15 minutes. Following the meal we will take further blood samples (from the cannula and finger pricks) for the next 15, 30, 45, 60, 90, 120, 150 and180 minutes. The amount of blood that will be collected at every time point will be about1.2 teaspoon of blood (approximately 6 mL).At the same time intervals the subjects will be instructed to fill in visual analogue scales on feelings of fullness, hunger, desire to eat and prospective food consumption.Visual analogue scales are 100 mm continuous lines anchored with opposing answers to a specific question asked. The specific questions asked will be, 'How hungry do you feel?', 'How full do you feel?', 'How strong is your desire to eat?', ' How much more food do you think you can eat?'. The subjects will be instructed to make a mark on the line which corresponds with their subjective feeling. After 3 hours, the cannula will be removed and the subjects will be instructed to an ad libitum lunch. After finish the lunch, the subjects will also be asked to complete a visual analogue scales (VAS) for the measurement of hunger and feelings of fullness. After which,subjects are free to leave Clinical Nutrition Research Centre. During the entire testing period the subjects will be instructed to remain rested and in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Age between 21-40 years
* Weight of at least 45 kg
* Body mass index between 18 to 25 kg/m2
* Normal blood pressure (≤140/90 mmHg)
* Fasting blood glucose <6.0 mmol/L

Exclusion Criteria:

* Are a female who is pregnant
* Partake in sports at the competitive and/or endurance levels
* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Have major chronic disease such as heart disease, cancer or diabetes mellitus
* Take insulin or drugs known to affect glucose metabolism
* Intentionally restrict food intake
* Have major medical or surgical event requiring hospitalization within the preceding 3 months
* Have taken antibiotics for 3 months before the study period
* Are a smoker
* Are an overnight shift worker
* Have any known food allergy (example anaphylaxis to peanuts)
* Having active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV).
* Are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC
* Have poor veins impeding venous access
* Have any history of severe vasovagal syncope blackouts or near faints following blood draws

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
glycemic response | up to 180 minutes
  using Hemocue analyzer
Insulin response | up to 180 minutes
  using COBAS Analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

REFERENCES:
- [Derived] Sun L, Goh HJ, Govindharajulu P, Leow MK, Henry CJ. Postprandial glucose, insulin and incretin responses differ by test meal macronutrient ingestion sequence (PATTERN study). Clin Nutr. 2020 Mar;39(3):950-957. doi: 10.1016/j.clnu.2019.04.001. Epub 2019 Apr 27. PMID 31053510